CLINICAL TRIAL: NCT05904873
Title: Can a Preoperative Cold Press Test be a Predictor of Pain After Third Molar Surgery?
Brief Title: Cold Press Test and Post Operative Pain Relationship
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinem Büşra Kıraç Can (Other)
Responsible Party: Sponsor-Investigator, Sinem Büşra Kıraç Can, DDS, PhD, Marmara University
Organization: Marmara University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: coldprsstst
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Post-operative Pain, Acute; Pain Threshold
Keywords: Cold Pressor Test; Post-operative Pain; Mandibular Third Molar
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The researcher who performs the ice test and the researcher who performs the surgical procedures are different from each other. The researcher performing the surgical procedure cannot know the ice test results of the participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The group who removed their hands from ice packs before 240 seconds (Experimental): In our study, a cold pressor test was applied to the participants in order to measure the pain tolerance according to the time duration they could keep their hands on the ice pack before the operation. Participants were prepared for an ice test in another area other than the operation area. Participants were asked to place their hands on standardized ice packs and keep them on the ice pack for 240 seconds. It was also said that if they could not tolerate pain, they could remove their hands from the ice before 240 seconds. The participants were asked to express the pain as a number between 0 (no pain) and 10 (unbearable pain) according to the visual analog scale when they removed their hands from the ice pack. Participants were divided into two groups according to the time duration of ice test as less than 240 seconds and equal to seconds.
  Interventions: Procedure: Mandibular Third Molar Surgery
- The group that can keep their hands on ice packs for 240 seconds (Experimental): In our study, a cold pressor test was applied to the participants in order to measure the pain tolerance according to the time duration they could keep their hands on the ice pack before the operation. Participants were prepared for an ice test in another area other than the operation area. Participants were asked to place their hands on standardized ice packs and keep them on the ice pack for 240 seconds. It was also said that if they could not tolerate pain, they could remove their hands from the ice before 240 seconds. The participants were asked to express the pain as a number between 0 (no pain) and 10 (unbearable pain) according to the visual analog scale when they removed their hands from the ice pack. Participants were divided into two groups according to the time duration of ice test as less than 240 seconds and equal to 240 seconds.
  Interventions: Procedure: Mandibular Third Molar Surgery

INTERVENTIONS:
Procedure: Mandibular Third Molar Surgery — All surgical procedures were carried out by a single dental(maxillofacial) surgeon different from the clinician performing the cold testing. A total of 4 cc of local anesthetic solution containing 40 mg/ml articaine and 0.005 mg/ml epinephrine was applied to the inferior alveolar and buccal nerve blocks before the surgical procedure. In all cases, the mucoperiosteal flap was raised and bone was removed from the buccal and distal parts of the impacted tooth with burs, while protecting the papilla between the first and second molars during flap design. Before extraction, if necessary, the third molar was divided and tooth extraction was performed with elevators. The flap was brought to its original position and closed with silk suture material.

SUMMARY:
The goal of this clinical trial is to investigate whether it is possible to get a preliminary idea about the postoperative pain in the patient with the results of a practical cold press test applied to American Society of Anesthesiologists(ASA) 1 and 2, healthy, male patients aged 16-35 before extraction of the lower third molar. The main question it aims to answer are:

• Can post-operative pain be predicted with an cold test that can be applied more practically than conventional quantitative sensory tests applied preoperatively? Participants will need to keep their hands on ice for 240 seconds prior to third molar surgery. When they take their hands off the ice, they will be asked to describe their pain on the visual analog scale. After the operation, the participants are required to mark whether they use painkillers every 8 hours in their pain follow-up forms and the pain they feel according to the visual analog scale.

Depending on the endurance time of the participants to keep their hands on the ice; Two different groups were determined as less than 240 sec and equal to 240 sec. The pain scores and the amount of painkiller use between these two groups were compared with each other.

ELIGIBILITY:
Inclusion Criteria:

* The impacted third molar should be class 1 or 2 and position B according to Pell & Gregory classification.
* The impacted third molar should be asymptomatic.
* The impacted third molar should be located in the mandible and be in the mesioangular or vertical position.
* To be male gender
* To be in American Society of Anesthesiologists 1 or 2 classification
* To be between the ages of 16-35

Exclusion Criteria:

* Intolerance to non-steroidal anti-inflammatory drugs
* Smoking more than 10 cigarettes a day
* Operation time exceeding 20 minutes
* Individuals who have performed third molar tooth extraction

Ages: 16 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Gonadal hormones are hypothesized to contribute to greater clinical and experimental pain experience in female patients compared to male patients. Therefore, the study group consisted of male patients only.
Enrollment: 30 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Measurement of Post-Operative Pain | 4 days
  To measure postoperative pain, all participants were given a form to fill out after surgery. In the form, there were areas where the participant should indicate pain between 0 and 10 according to the VAS scale . Forms were collected from each participant at the end of 4 days after the operation.

SECONDARY OUTCOMES:
Measurement of Painkiller Use In The Post Operative Period | 4 days
  To measure the amount of painkillers used post-surgery, all participants were given a form to fill out. In the form, there were areas where the participant should mark the use of ibuprofen in the first 0-2 hours and then every 8 hours. If paracetamol, which is the rescue medicine, is used, it was requested to mark the time and date in the table in the last part of the form. Forms were collected from each participant at the end of 4 days after the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Sinem Busra Kirac Can, Principal Investigator — Marmara University; Gülcan Berkel, Asist Prof, Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)